CLINICAL TRIAL: NCT05872256
Title: A Demonstration of the Hair and Scalp Benefits of 0.045% Tazarotene/0.01% Halobetasol Lotion in Scalp Psoriasis
Brief Title: A Demonstration of the Hair and Scalp Benefits of Duobrii in Scalp Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dermatology Consulting Services, PLLC (Network)
Collaborators: Ortho Dermatologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCS-165-22
Record Dates: First submitted 2023-05-14; First posted 2023-05-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Scalp Psoriasis

STUDY DESIGN:
Intervention Model Description: All subjects will receive the currently marketed and FDA approved Duobrii lotion to the scalp for the treatment of scalp psoriasis.
Masking Description: All subjects will receive Duobrii lotion for scalp application to all areas afflicted with scalp psoriasis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active Arm (Other): 0.045% Tazarotene/0.01% Habetasol Lotion apply once daily at bedtime to the scalp afflicted with psoriasis
  Interventions: Drug: 0.045% Tazarotene/0.01% Halobetasol Lotion

INTERVENTIONS:
Drug: 0.045% Tazarotene/0.01% Halobetasol Lotion — FDA approved drug for psoriasis treatment
  Other Names: Duobrii Lotion

SUMMARY:
The objectives of this research are to demonstrate the following:1. To demonstrate improvement in hair growth and hair appearance following 12 weeks of once daily treatment with tazarotene/halobetasol lotion in patients with moderate to severe scalp psoriasis.2. To demonstrate improvement in scalp itch reduction following 12 weeks of once daily treatment with tazarotene/halobetasol lotion in patients with moderate to severe scalp psoriasis.3. To pictorially demonstrate improvement in moderate to severe scalp psoriasis with 12 weeks of once daily treatment with tazarotene/halobetasol lotion.4. To assessment patient perceptions of the value of a lotion in the treatment of moderate to severe scalp psoriasis.

DETAILED DESCRIPTION:
Male or female subjects with moderate to severe scalp psoriasis will present to the research center for evaluation for study entry. They will have been advised to present to the research center with clean hair and no topical products applied to the scalp. If found to be suitable by meeting all inclusion criteria and none of the exclusion criteria, subjects will undergo scalp psoriasis evaluation by the dermatologist investigator for erythema, scaling, and induration. The subjects will also assess each plaque for redness, thickness, and scaling. The subjects and the dermatologist will assess the hair for lack of hair shine, poor manageability, frizziness, poor hair color, poor hair growth, and damaged cuticle structure. The subjects will assess scalp itch. Finally, digital photography will be conducted of the scalp psoriasis.Each subject will be dispensed one tube of tazarotene/halobetasol lotion for application to scalp once daily. Subjects will be provided with a diary. Subjects will be instructed to return to the research center in 4 weeks. A reminder text for compliance will be provided prior to the week 4 visit and for all return visits.Subjects will return to the research center at week 4 and week 8 and week 12 for the same assessments. At week 12, a consumer perception survey will also be administered. All diaries will be collected at week 12. Subjects will be allowed to keep any unused study product. Subjects will complete their study participation at week 12.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males or non-pregnant females 18+ years of age. 2. Plaque type moderate to severe scalp psoriasis suitable for topical treatment.

  3. Subjects must be in general good health as determined from a medical history.

  4. Subjects must read and sign the informed consent form after the nature of the study has been fully explained.

Exclusion Criteria:

* 1. Subjects with known allergies or sensitivities to ingredients contained in the test products.

  2. Subjects with pustular or erythrodermic psoriasis. 3. Subjects who are pregnant or nursing or planning to become pregnant during the course of the study.

  4. Subjects who are currently participating in any other clinical study (i.e., dermal patch, use tests, investigational drug or devices, etc.).

  5. Subjects viewed by the investigator as not being able to complete the study. 6. Subjects using any type of lotion, medication, or other topical product to the scalp psoriasis within 2 weeks of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Hair Growth | 12 weeks
  Improvement in hair growth due to scalp psoriasis treatment
Scalp Itch | 12 weeks
  Reduction in scalp itch due to scalp psoriasis treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zoe D Draelos, MD, Principal Investigator — Dermatology Consulting Services, PLLC
Locations (1):
- Dermatology Consulting Services, PLLC, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The data will not be shared.